CLINICAL TRIAL: NCT07356986
Title: Stelo Real-time Continuous Glucose Monitor Use Postpartum for Lifelong Optimal Wellness
Acronym: STELO-GLOW
Status: Not yet recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: DexCom, Inc. (Industry); University of Pennsylvania (Other); Sansum Diabetes Research Institute (Other)
Responsible Party: Principal Investigator, Amy Miyoshi Valent, Principal Investigator, Oregon Health and Science University
Other Study IDs: STUDY00028947
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Gestational Diabetes; Postpartum
Keywords: Continuous Glucose Monitoring; Postpartum Glucose Management
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postpartum Stelo Users: Postpartum individuals with their most recent pregnancy complicated by Gestational Diabetes Mellitus (GDM)
  Interventions: Device: Dexcom Stelo real-time Continuous Glucose Monitor

INTERVENTIONS:
Device: Dexcom Stelo real-time Continuous Glucose Monitor — The Stelo Glucose Biosensor is an over-the-counter integrated Continuous Glucose Monitor (iCGM) intended to continuously measure, record, analyze, and display glucose values in people 18 years and older not on insulin. Participants will use Stelo for the 6 weeks following delivery and for 15 days at 3 months, 6 months, 9 months, and 1 year postpartum.

SUMMARY:
The purpose of this prospective observational study is to gather exploratory and practical use data of the Dexcom Stelo Glucose Biosensing System (Stelo), an over-the-counter (OTC) real-time Continuous Glucose Monitoring (CGM) system among patients with Gestational Diabetes Mellitus (GDM) in their most recent pregnancy.

DETAILED DESCRIPTION:
50 postpartum individuals with GDM during their most recent pregnancy will be enrolled in this prospective observational study. In a prior study looking at real-world use of Dexcom G7 CGM during pregnancy among people with GDM, feasibility was demonstrated as well as a willingness to continue CGM use during the postpartum period.

Each enrolled subject will be asked to train and wear the Dexcom Stelo glucose biosensor system continuously for the first 6 weeks after delivery and at least 1 sensor wear every 3 months (up to 15 days at 3, 6, 9, and 12 months) for the remainder of the postpartum period up to 1 year from delivery. The first insertion will be performed under trained observation and additional supplies will be provided every 3 months. Participants will be trained and instructed to enter meals, activity, lactation, and anti-diabetic medications (if applicable) in the Dexcom Stelo App as they are willing to input. Subjects will be provided education on the importance of nutrition, physical activity, and mental health in postpartum and long-term health and tips on how to use CGM data to encourage lifestyle and behavioral modifications.

ELIGIBILITY:
Inclusion Criteria:

* Gestational Diabetes Mellitus (GDM) diagnosis by 1- or 2-step Oral Glucose Tolerance Test (OGTT) during pregnancy or >= 200 mg following any glucose challenge (50g, 75g, 100g)
* Has a smart phone compatible to support Dexcom Stelo app
* Able to read, write, and understand English
* Meet Stelo Glucose Biosensor Indications for Use (IFU) per approved commercial labeling
* Willing to follow all study procedures

Exclusion Criteria:

* Greater than 6 weeks and 6 days postpartum at enrollment
* Preexisting Type 1 Diabetes (T1D) or Type 2 Diabetes (T2D)
* End-stage renal failure (on dialysis)
* Heart failure
* Other uncontrolled high-risk condition as determined exclusionary by site investigators
* Extensive skin changes/diseases that preclude wearing the required system on normal skin (e.g. extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis) at the proposed wear sites
* Known severe allergy to medical-grade adhesives
* Any condition that, in the opinion of the investigator, would interfere with their participation in the trial
* Obesity surgery
* Insulin use prior to discharge home from the delivery admission
* Current participation in another postpartum Continuous Glucose Monitoring (CGM) or lifestyle intervention trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postpartum individuals with pregnancies complicated by GDM.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Mean Glucose | Measured from birth to 6 weeks postpartum, and for 15 days at 3, 6, 9, and 12 months postpartum.
  24-hour mean glucose based on Stelo Glucose Biosensor readings
Glucose Percent Time in Range | Measured from birth to 6 weeks postpartum, and for 15 days at 3, 6, 9, and 12 months postpartum.
  Percent time-in-range (percent of the time between 70-140 mg/dL or 70-120 mg/dL) based on Stelo Glucose Biosensor readings
Glucose Percent Time Above Range | Measured from birth to 6 weeks postpartum, and for 15 days at 3, 6, 9, and 12 months postpartum.
  Percent time-above-range (percent of the time above 140 mg/dL or 120 mg/dL) based on Stelo Glucose Biosensor readings
Postpartum Fasting Glucose | Measured at 6 and 12 months postpartum
  Postpartum fasting glucose as determined by a blood test
Postpartum A1C | Measured at 6 and 12 months postpartum
  Postpartum Hemoglobin A1C as determined by a blood test

CONTACTS AND LOCATIONS:
Overall Officials: Amy M Valent, DO, MCR, Principal Investigator — Oregon Health and Science University; Celeste Durnwald, MD, Principal Investigator — University of Pennsylvania; Kristin Castorino, DO, Principal Investigator — Sansum Diabetes Research Institute
Locations (3):
- United States (3):
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon request following publication.